CLINICAL TRIAL: NCT03772340
Title: Motion Sifnos: A Randomized, Double-blind, Placebo-controlled Study to Investigate the Efficacy of Tradipitant in Subjects Affected by Motion Sickness During Travel
Brief Title: Motion Sifnos: A Study to Investigate the Efficacy of Tradipitant in Subjects Affected by Motion Sickness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VLY-686-2401
Record Dates: First submitted 2018-11-28; First posted 2018-12-11 (Actual); Results first posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-04

CONDITIONS: Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tradipitant (Experimental)
  Interventions: Drug: Tradipitant
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tradipitant — Oral capsule
  Arms: Tradipitant
Drug: Placebo — Oral capsule
  Arms: Placebo

SUMMARY:
Randomized, double-blind, placebo-controlled investigating the efficacy of tradipitant in the treatment of motion sickness.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female patients aged 18 - 75 years (inclusive);
* Body Mass Index (BMI) of ≥18 and <40 kg/m2;
* History or symptoms consistent with motion sickness

Exclusion Criteria:

* Chronic nausea due to condition other than motion sickness;
* A positive test for drugs of abuse at the screening or evaluation visits;
* Clinically significant deviation from normal clinical laboratory results

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-06-06 (Actual); Study Completion 2019-06-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanda Investigational Site, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://www.frontiersin.org/articles/10.3389/fneur.2020.563373/full

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tradipitant | Placebo
Started | 63 | 63
Completed | 63 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tradipitant | Placebo | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.6 (11.44) | 39.7 (12.65) | 39.1 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 97
  Male | 13 | 16 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 21 | 43
  Not Hispanic or Latino | 41 | 42 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 1 | 1
  Asian | 6 | 8 | 14
  Black or African American | 6 | 4 | 10
  Native Hawaiian or Pacific Islander | 2 | 0 | 2
  White | 44 | 49 | 93
  Other | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 63 | 63 | 126
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.58 (5.03) | 27.87 (4.858) | 27.22 (4.967)

OUTCOME MEASURES:

1. Primary Outcome: The Most Severe Motion Sickness Severity During Vehicle Travel
Description: As measured by the Motion Sickness Severity Scale (MSSS) (NRS 0-6); Lower score indicates improvement
Time Frame: 1 day
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 63 | 63
units on a scale | 3.4 (0.238) | 3.75 (0.239)

2. Primary Outcome: Percentage of Vomiting
Description: Defined as subjects ever vomited (MSSS=6) or terminated early due to severity during the vehicle travel. As measured by the Motion Sickness Severity Scale (NRS 0-6).
Time Frame: 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Tradipitant | Placebo
Number analyzed (Participants) | 63 | 63
Participants
  Vomiting No | 52 | 38
  Vomiting Yes | 11 | 25

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) were collected from the time of the subject's informed consent signature until the end of the subject's study participation. AEs reported or learned up to 7 days after the subject's last study visit or a new SAE(s) up to 30 days after last study visit were recorded. AEs were monitored for approximately one month after randomization.
Arm/Group | Tradipitant | Placebo
All-Cause Mortality (participants affected / at risk) | 0/63 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/63
Other Adverse Events (participants affected / at risk) | 39/63 | 39/63
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tradipitant (N=63) | Placebo (N=63)
Motion Sickness (Ear and labyrinth disorders) | 19 | 27
Somnolence (Nervous system disorders) | 17 | 8
Headache (Nervous system disorders) | 8 | 5
Nausea (Gastrointestinal disorders) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/40/NCT03772340/Prot_SAP_000.pdf